CLINICAL TRIAL: NCT05649995
Title: Effectiveness of Pain Science Education in People With Symptomatic Knee Osteoarthritis: A Randomized Controlled Study
Brief Title: Effectiveness of Pain Science Education in People With Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Hilal Ata Tay, Principal investigator, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 092022160
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; pain; knee; education
MeSH Terms: conditions — Osteoarthritis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain science education group (Experimental): the program integrated with pain science education (exercise, walking program and recommendations for reducing sedentary behaviors)
  Interventions: Other: Pain science education driven physiotherapy program
- Biomedical education group (Experimental): the program integrated with biomedical education (exercise, walking program and recommendations for reducing sedentary behaviors)
  Interventions: Other: Biomedical education driven physiotherapy program

INTERVENTIONS:
Other: Pain science education driven physiotherapy program — Pain science training will be carried out as described by Moseley and Butler. Topics covered within the scope of pain science education are planned to include: neurophysiology of pain, synapses, peripheral sensitization, central sensitization, plasticity of the nervous system. The aim of the training will be to teach participants that pain is a multifactorial experience rather than just tissue injury. Participants in this group will be told about the importance of physical activity integrated with pain science education (i.e., explaining that physical activity is the key to bioplasticity and causing changes in our system) and why sedentary behaviors should be reduced (reducing sedentary behaviors reduces the overprotectiveness of the pain system).
  Arms: Pain science education group
Other: Biomedical education driven physiotherapy program — Participants in this group will be planned to increase their knowledge of knee anatomy, knowledge of knee OA and knee OA risk factors, and the importance of increasing physical activity and reducing sedentary behavior in reducing osteoarthritic pain and improving overall health. The importance of physical activity by integrating it with biomedical education (as physical activity can help strengthen muscles, protect joint function, and improve sleep and general health) and the necessity of reducing sedentary behaviors will be discussed within the framework of biomedical education.The main difference of standard education from pain science education will be that it does not contain information about pain mechanisms mentioned in pain science education.
  Arms: Biomedical education group

SUMMARY:
The aim of this study is to determine the effectiveness of the program integrated with pain science education for people with painful knee osteoarthritis (OA). Another purpose of the study is to evaluate whether the program integrated with pain science education is more effective than the program integrated with biomedical education.

DETAILED DESCRIPTION:
Contemporary pain science education provides a scientific basis for the increased sensitivity produced in chronic pain due to adaptations in the central nervous system. In the literature, pain science education has been shown to reduce unhelpful pain beliefs and improve pain, function, and disability in several chronic musculoskeletal pain states, but data specific to knee OA are lacking.

Patients with knee osteoarthritis who meet the inclusion criteria and agree to participate in the study will be included. The participants will be randomly divided into two groups. These groups are: a) intervention group, where the program integrated with pain science education and b)control group, where the program integrated with biomedical education.

Three weeks of face-to-face sessions in both groups will be followed by three weeks of telerehabilitation sessions. Telerehabilitation sessions will be applied as phone calls or video conference sessions, according to the participant's request. All sessions will be conducted one-on-one.

Face-to-face sessions for both groups:

* 3 sessions in total,
* 1 day a week for 3 weeks,
* Each session will last approximately 60 minutes for the control group and the intervention group.
* Each face-to-face session will include education and physiotherapy program. Biomedical education for the control group and pain science education for the intervention group will be applied. Visuals and presentations will be used in the education of both groups. The presentations and visuals that will be used in pain science education and biomedical education will be different. The physiotherapy program will be the same for both groups. Physiotherapy program will be applied after education in both groups. In the physiotherapy program, all participants will be given knee exercises and will be asked to take a walk twice a week as homework and suggestions will be made to reduce their sedentary behavior. The exercises given to both groups will be the same.

Telerehabilitation sessions for both groups:

* 3 sessions in total,
* 1 day a week for 3 weeks,
* Each session is approximately 15-20 minutes,
* Each session will include education, recommendations (especially about increasing physical activity and reducing sedentary behaviour), answering questions if any, and discussion.

The homework and suggestions to be given to the participants in the intervention group will be integrated with the pain science education, while the homework and suggestions to be given to the participants in the control group will be integrated with the biomedical education. For example, it will be explained to a participant in the intervention group that walking will regulate increased sensitivity in the central nervous system and ensure plasticity (using stories, examples in a way that the participant can understand). It will be explained to the participant in the control group that walking will strengthen their muscles and will be beneficial for general health and joint health.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with knee osteoarthritis according to the criteria of the American College of Rheumatology (ACR).
* Being between the ages of 45-65
* Having knee pain lasting at least 6 months
* Average knee pain intensity of ≥4 on 11- point numeric rating scale in the past week
* Having Turkish as mother tongue
* Being literate

Exclusion Criteria:

* Having health problems (eg heart or lung disease) that prevent safe participation in physical activity interventions as listed in the American College of Sports Medicine Guidelines.
* Neurological disorders affecting the lower extremity (eg multiple sclerosis or stroke)
* Using an assistive device
* Being diagnosed with OA in joint areas other than the knee joint
* Presence of inflammatory arthritis (including rheumatoid arthritis)
* Presence of any condition that affects decision making/memory (eg Alzheimer's, dementia)
* Knee replacement/surgery planning for the next 3 months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions) T3 (within 7 week after the end of the telerehabilitation sessions)
  Assessed using the numeric rating scale that assesses pain intensity (range 0-10 and higher values are indicative of higher pain intensity)
Changes in pain frequency | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  Assessed using a closed question about knee pain frequency in the last week (How many times in the last week have you felt this pain?". The answer options are: Never, rarely (once a week) occasionally (2 to 3 times a week), often (more than 3 times a week) and always.
Changes in WOMAC (Western Ontario and McMaster Universities) index | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions) T3 (within 7 week after the end of the telerehabilitation sessions)
  womac will be used to assess pain, stiffness and physical function
Changes in the level of pain catastrophizing | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  Assessed using the Pain Catastrophizing Scale (range 0-52 and higher values are indicative of higher pain catastrophizing)

SECONDARY OUTCOMES:
Changes in fear of movement | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  assessed using the Tampa Scale of Kinesiophobia, which assesses fear of movement (range: 13-52 and higher values are indicative of higher levels of fear of movement)
Changes in health-related quality of life | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  assessed using the self-reported Short Form-12 questionnaire
Changes in physical activity level | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  assessed using the International Physical Activity Questionnaire (IPAQ) -Short Form.
Changes in sleep quality level | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  assessed using the Pittsburgh Sleep Quality Index (the higher score indicates worse sleep quality).
Changes in sedentary time and sedentary behavior | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions)
  The questions to be used in the evaluation of sedentary behaviors and sedentary time were adapted using the scale developed by Salmon (Salmon et al, 2003).
  The sedentary behaviors of the participants will be questioned for their activities in eight different categories. These activities include: watching television, using a computer, reading a book, surfing the Internet on the phone, engaging in arts & games & hobbies (e.g. playing chess, knitting, sewing, drawing), chatting or socializing, just doing nothing to rest, to travel by vehicles such as buses, cars.
Evaluation of Satisfaction Level from Pain Science Education | T1 (within 1 week after the end of the face-to-face sessions)
  Satisfaction will be measured through visual analogue scale 0-100mm (0= not satisfied at all; 100 = very satisfied).
Adherence to rehabilitation program | Baseline (T0, 1 week before beginning of the study); T1 (within 1 week after the end of the face-to-face sessions); T2 (within 1 week after the end of the telerehabilitation sessions) T3 (within 7 week after the end of the telerehabilitation sessions)
  Adherence to the walking program will be calculated by evaluating the duration and frequency of their walks each week.
  Adherence to the knee exercises will be calculated by evaluating the number of the days they exercise in each week.
  Adherence to recommendations about sedentary behavior will be calculated by evaluating the total time they sit and the frequency and duration of the breaks they take while sitting.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Ata Tay, Principal Investigator — Marmara University
Locations (2):
- Turkey (Türkiye) (2):
  - Marmara University, Istanbul, Maltepe
  - Marmara University Pendik Training and Research Hospital, Istanbul